CLINICAL TRIAL: NCT07251400
Title: The Analgesic Efficacy of Ultrasound-guided Erector Spinae and Rectus Sheath Block in Patients Undergoing Laparoscopic Inguinal Hernia Repair: a Randomized Controlled Trial
Brief Title: Analgesic Efficacy of Erector Spinae and Rectus Sheath Block in Patients Undergoing Laparoscopic Inguinal Hernia Repair
Acronym: analgesia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeliha Alicikus, assoc. prof. dr, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zeliha20
Record Dates: First submitted 2025-11-16; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Erector Spinae Plane Block; Laparoscopic Inguinal Hernia Repair
Keywords: postoperative analgesia; erector spinae plane block; inguinal hernia repair

STUDY DESIGN:
Intervention Model Description: * Group 1: ESB (n = 30)
  * Group 2: RSB (n = 30)
  * Group 3: LA infiltration (n = 30)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESB (Erector spinae plane block) group (Active Comparator): The ESP block will be applied under general anesthesia after skin closure lateral decubitus position. The ultrasound probe will be placed in a longitudinal parasagittal orientation approximately 3 cm lateral to the T7 spinous process. Using the inplane technique, a 22-gauge, 80 mm needle will be advanced craniocaudally, and 30 ml of 0.25% bupivacaine will be injected between the erector spinae muscle and the transverse process. ESPB will be performed bilaterally, with 30 ml of local anesthetic administered to the plane of the erector spinae on each side.
  Interventions: Procedure: Erector spinae plane block
- RSB (Bilateral rectus sheath block) group (Active Comparator): Before recovery from anesthesia, an ultrasound-guided rectus sheath block will be performed after the skin incision is closed. the rectus sheath and the posterior aspect of the rectus abdominis muscle an 80 mm, 22-gauge short-tapered needle will be advanced anterolaterally to medially using in-plane placement with real-time assessment, Once the tip is correctly positioned in the intended plane, 20 mL of a local anesthetic, typically bupivacaine at a concentration of 0.25%, will be administered on each side for effective analgesia.
  Interventions: Procedure: Erector spinae plane block
- LA infiltration group (Active Comparator): Patients who will receive local anesthesia only for surgical incisions will be considered the control group. 20 ml of 0.25% bupivacaine will be applied to the surgical incisions, and no plane block will be performed
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — postoperative analgesia for inguinal hernia repair
  Other Names: Bilateral rectus sheath block

SUMMARY:
The aim of this study was to compare the effectiveness of ultrasound-guided erector spinae plane block and rectus sheet block on postoperative pain in patients undergoing laparoscopic bilateral hernia repair.

DETAILED DESCRIPTION:
Multiple factors play a critical role in the development of pain after laparoscopic bilateral inguinal hernia repair surgery. These include parietal stimulation from the surgical incision, visceral stimulation from the peritoneum, and manipulation of intra-abdominal structures. Somatic innervation of the anterior abdominal wall is provided by the thoracolumbar spinal nerves T6-L1. Innervation of the skin above the umbilicus is provided by cutaneous nerves T6 to T9. The area around the umbilicus is innervated by T10, while the underlying skin is innervated by T11, T12, and L1. The peritoneum contains "silent nociceptors" that are activated by surgical injury and intraperitoneal inflammation and contribute to visceral pain. The neuro-immuno-humoral pain pathways involved in abdominal surgery involve somatic and autonomic nerves. Parasympathetic activation and decreased vagal tone have been shown to influence perioperative outcome because they exacerbate inflammation associated with gastrointestinal dysfunction. Thoracic epidural analgesia is still considered the gold standard for postoperative analgesia in major abdominal surgery; however, concerns about the risk of major complications such as hypotension, motor block, epidural hematoma, and abscess sometimes limit its use. Intravenous morphine administration is a cornerstone of pain management, but the side effects seen after opioid use limit its use. An ideal multimodal analgesic method includes regional blocks (neuraxial blocks [epidural and paravertebral analgesia], plane blocks [transversus abdominis plane blocks and rectus sheath block], intravenous analgesic medications (nonsteroidal anti-inflammatory drugs, cyclooxygenase-2 selective inhibitors, or single intraoperative dexamethasone), and surgical field infiltration.

Erector spinae plane block (ESPB) was first described for the treatment of thoracic neuropathic pain and has since become an effective periparavertebral regional anesthesia technique applied to prevent postoperative pain in various surgeries. ESPB was initially applied at the T5 level, but more recently has been shown to be effective in providing comprehensive somatic and visceral abdominal analgesia when applied at the T7-T9 level. It is easier to administer than thoracic epidural anesthesia and thoracic paravertebral block. The effectiveness of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy has been studied. A study evaluating ESPB with bilateral ultrasound concluded that it provides effective analgesia in patients and significantly reduces analgesia requirements, extending to up to 1 week. Bilateral rectus sheath block (RSB) provides analgesia to the anteromedial abdominal wall and periumbilical area by blocking spinal dermatomes T9, T10, and T11. RSB provides analgesia to the anterior cutaneous branches of the intercostal nerves and is therefore well-suited for postoperative analgesia for midline abdominal incisions. Although initially developed to provide anterior abdominal muscle relaxation, RSB has subsequently been used for pain relief after abdominal surgery. This fascial plane block involves the deposition of a local anesthetic between the rectus muscle and the posterior sheath to anesthetize the terminal branches of the lower thoracic spinal nerves T7-T12. A recent meta-analysis of 698 patients found that RSB improved pain control and reduced opioid consumption for up to 12 hours postoperatively, with no significant adverse events reported.

The primary objective of this study was to compare the effectiveness of ultrasound-guided erector spinae plane block and rectus sheet block on postoperative pain in patients undergoing laparoscopic bilateral hernia repair. The secondary objective was to compare opioid consumption in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and under 70 years of age
* ASA I-III

Exclusion Criteria:

* Patients with ASA IV,
* known neurological or psychiatric disorders,
* asthma or COPD,
* long-term drug or alcohol abuse,
* diabetes mellitus,
* BMI >35,
* intellectual disability,
* contraindications for EPSP or RSB,
* massive bleeding, coagulopathy
* those with significant systemic conditions undergoing emergency surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
postoperative pain in patients undergoing laparoscopic bilateral hernia repair | 24 hours after extubation
  VAS score

SECONDARY OUTCOMES:
Total Postoperative Opioid Consumption | immediately after the surgery
  remifentanyl

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Alıcıkuş, asc prof, Principal Investigator — Umraniye ERH
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No